CLINICAL TRIAL: NCT02650570
Title: Mitochondrial Respiratory Function in Mammalian Skeletal Muscle: Metabolic Insights Into Cancer and Burn Cachexia Through Comparative Physiology of Humans and Marine Mammals
Brief Title: Mitochondrial Respiratory Function in Mammalian Skeletal Muscle
Status: Terminated | Type: Observational
Why Stopped: Funding Ended
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0056
Record Dates: First submitted 2015-12-08; First posted 2016-01-08 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cancer; Cachexia
Keywords: Cancer; Cachexia
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma will be collected and retained in the PI lab.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Head/Neck Cancer: Subjects diagnosed with advanced (stages III or IV), persistent (recurrence within 6 months) or recurrent head and neck squamous cell carcinoma (HNSCC)
- Healthy Control: Healthy controls age matched to the Head/Neck cancer group.

SUMMARY:
The purpose of this study is to determine whether skeletal muscle mitochondrial function is altered in patients with head and neck cancer compared to healthy controls.

DETAILED DESCRIPTION:
20 men and women, 30-60 years, equally divided between patients diagnosed with advanced (stages III or IV), persistent (recurrence within 6 months) or recurrent head and neck squamous cell carcinoma (HNSCC) (n=10) and healthy age matched control subjects (n=10) will be studied.

Muscle biopsies will be collected from cancer patients before and after a 4 week standard of care (SOC) treatment. Muscle biopsies from healthy control subjects will be collected at baseline only.

Lean body mass and fat mass will be determined by a DEXA scan before and after 4 week SOC treatment (cancer patients) to document any change in body composition (cachexia), and at baseline only in the age-matched healthy controls.

Blood will be collected from both cancer patients and healthy subjects to examine hormone levels at the time of biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 30-60 years.
2. Diagnosed with advanced (stages III or IV), persistent (recurrence within 6 months) or recurrent head and neck squamous cell carcinoma (HNSCC) and being treated at UTMB (n=10).
3. Healthy sex and age matched controls (n=10.)
4. Able to comprehend risks and sign a consent form.
5. Fluent in English

Exclusion Criteria:

1. Significant renal or heart disease or any acute metabolic disease.
2. Evidence of hepatitis as indicated by a 3-fold increase in of 2 out of 3 liver enzymes.
3. Diabetes mellitus or other untreated endocrine disease.
4. Recent (within 3 months) treatment with anabolic steroids.
5. Ongoing anticoagulant therapy.
6. Polycystic ovary syndrome (PCOS) and/or hyperthecosis.
7. Non-classical adrenal hyperplasia.
8. Cushing's syndrome.
9. Pregnancy.
10. Hyperprolactinoma, hypothyroidism.
11. Granulocyte Count below 1.5x103/µL
12. Platelet Count below 150 x 103/µL
13. White Blood Cell Count below 1.0x103/µL
14. Hemoglobin below 8.0 g/dL
15. Organ transplant, HIV, or other criteria deemed immunosuppressing by the PI or study physician.
16. Any other circumstance deemed exclusionary by the PI or study physician.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects diagnosed with advanced (stages III or IV), persistent (recurrence within 6 months) or recurrent head and neck squamous cell carcinoma (HNSCC) (n=10).
  Healthy Controls (n=10).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Baseline skeletal muscle oxygen consumption (pmol O2/s*mg) in head and neck cancer patients and healthy age-matched controls | Baseline
  Aerobic respiration will be measured from skeletal muscle biopsies of the vastus lateralis using Oroboros O2K high resolution respirometry. The average maximal skeletal muscle oxygen consumption of 10 head and neck cancer subjects will be compared to the average of 10 healthy controls.
Skeletal muscle oxygen consumption (pmol O2/s*mg) in head and neck cancer patients following 4 weeks of standard of care. | 4 weeks
  Aerobic respiration will be measured from skeletal muscle biopsies of the vastus lateralis using Oroboros O2K high resolution respirometry. The average maximal skeletal muscle oxygen consumption of 10 head and neck cancer subjects after 4 weeks of standard of care (including chemotherapy, corticosteroids, etc. as prescribed by physician) will be compared to the average of their baseline measures.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No